CLINICAL TRIAL: NCT05116813
Title: An Open-label Safety Study of Dipraglurant (ADX48621) in Patients With Parkinson's Disease Receiving Levodopa-based Therapy With or Without Concomitant Dopaminergic Medications
Brief Title: Open-label Safety Study of Dipraglurant (ADX48621) in Patients With Parkinson's Disease Receiving Levodopa-based Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated prior to completing enrollment goals due to COVID-related difficulties in recruiting patients
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADX48621-302
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias
Keywords: Parkinson's disease; Dyskinesia; Levodopa-induced Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias | interventions — 6-fluoro-2-(4-(pyridin-2-yl)but-3-yn-1-yl)imidazo(1,2-a)pyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dipraglurant TID (Experimental)
  Interventions: Drug: Dipraglurant

INTERVENTIONS:
Drug: Dipraglurant — Oral 50 mg and 100 mg tablet
  Other Names: ADX48621

SUMMARY:
This open-label study is designed to assess the long-term safety and tolerability of dipraglurant in PD patients for up to 52 weeks (at doses of 150-300 mg per day) for patients that have completed an Addex sponsored double-blind clinical trial of dipraglurant.

ELIGIBILITY:
Inclusion Criteria:

* Completed an Addex randomized controlled study of dipraglurant and, in the judgement of the Investigator, may benefit from open-label treatment
* Able to take study drug 3 times daily and no less than 3 hours apart
* Must be taking levodopa not less than 3 times daily throughout the study
* Must maintain stable regimen of antiparkinson's medications (including levodopa) and be willing to continue the same doses and regimens for the first 4 weeks of the study

Exclusion Criteria:

* Patient is judged by the Investigator to be inappropriate for the study (for reasons such as, but not limited to, significant noncompliance in the Addex randomized controlled study of dipraglurant)
* Use of amantadine or amantadine ER throughout the study
* Use of memantine throughout the study
* Any use of marijuana or other cannabis/cannabinoid products for the first 4 weeks of study participation

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability of dipraglurant as measured by incidence of adverse events | Baseline (Day 1) to Week 52
  Testing the safety and tolerability of dipraglurant in patients with Parkinson's Disease Levodopa-induced dyskinesia based on the incidence of adverse events reported by patients and/or as identified by the Investigator based on clinical assessments conducted during the study.

SECONDARY OUTCOMES:
Evaluate the continued utility of dipraglurant on dyskinesia as assessed by a change-from-baseline score on the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). | Baseline (Day 1) to Week 52
  The MDS-UPDRS is a Parkinson's Disease (PD) rating scale scored from 0-272; it evaluates progression of disease in patients with PD. A higher score indicates more severe PD.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Augusta University, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Rutgers, the State University of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Abington Neurologic Associates, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No